CLINICAL TRIAL: NCT03239496
Title: A Phase 3, Open-label, Multicenter Randomized Trial to Evaluate Humoral Immunogenicity of Various Schedules of Intramuscular Full-Dose and Intradermal Fractional Dose of Inactivated Polio Vaccine in Latin American Infants
Brief Title: A Study to Evaluate Immunogenicity of Intramuscular Full-Dose and Intradermal Fractional Dose of IPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV004
Record Dates: First submitted 2017-07-28; First posted 2017-08-04 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): 3 doses IPV IM at 10, 14 & 36 weeks of age incl. blood sampling at 10, 14, 18 & 40 weeks.
  Interventions: Biological: IPV
- Group B (Experimental): 2 doses IPV IM at 14 & 36 weeks of age incl. blood sampling at 14, 18, 36 & 40 weeks.
  Interventions: Biological: IPV
- Group C (Experimental): 3 doses f-IPV ID at 10, 14 & 36 weeks of age incl. blood sampling at 10, 14, 18 & 40 weeks.
  Interventions: Biological: f-IPV
- Group D (Experimental): 2 doses f-IPV ID at 14 & 36 weeks of age incl. blood sampling at 14, 18, 36 & 40 weeks.
  Interventions: Biological: f-IPV

INTERVENTIONS:
Biological: IPV — Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
  Arms: Group A; Group B
Biological: f-IPV — Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
  Arms: Group C; Group D

SUMMARY:
The study will assess and compare the immune response to full-dose inactivated polio vaccines (IPV) via intramuscular (IM) administration and of the fractional dose of inactivated poliovirus vaccine (f-IPV) via intradermal (ID) administration, in different schedule combinations in the Expanded Program on Immunization (EPI) primary series.

DETAILED DESCRIPTION:
This study prioritizes comparisons involving two-dose regimens recently recommended by the World Health Organization (WHO) Strategic Advisory Group of Experts on immunization (SAGE) and Pan American Health Organization (PAHO) in response to global IPV supply shortages 21. Furthermore, the study will provide data on the comparative humoral immunogenicity of various schedules to inform polio immunization policy for the post-eradication era.

The study population will include infants in Dominican Republic and Panama. Absence of wild and circulating vaccine derived polioviruses along with the lack of regular Supplementary Immunization Activities (SIAs) in the Latin America region provide an ideal epidemiologic setting to study polio vaccine immunogenicity.

Infants will receive two or three doses of full-dose IPV IM or f-IPV ID, in two schedules (10, 14 and 36 weeks and 14 and 36 weeks). Immunological and safety assessments will be made after one dose, two doses and three doses.

A total of 773 infants will be enrolled and distributed into 4 groups, according to a randomization scheme. During the study period, infants will be administered other concomitant vaccines according to the national schedules of the participating countries, but the effect, if any, of the concomitant administration on IPV immunogenicity will not be assessed.

Optimum immunogenicity expected from the dose(s) of IPV in the post-eradication era will have to be balanced with the cost and supply constraints of IPV. This study will be critical to determine how many doses of IPV and which schedule are optimal for the post-eradication era after the global cessation of Oral Polio Vaccine (OPV) use.

ELIGIBILITY:
Inclusion Criteria:

1. Infants of 6 weeks of age (-7 to + 7 days) on date of enrollment.
2. Healthy, as assessed from medical history and physical examination by a study physician,
3. Written informed consent obtained from parents or legal representatives who have been properly informed about the study and are able to comply with planned study procedures.

Exclusion Criteria:

1. Vaccinated with any poliovirus vaccine prior to inclusion,
2. A household contact with OPV vaccination history in the past 4 weeks,
3. HIV infection or pharmacologic immunosuppression,
4. Known allergy to any component of the study vaccines (phenoxyethanol, formaldehyde),
5. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular and intradermal injections,
6. Acute severe febrile illness on day of vaccination deemed by the Investigator(s) to be a contraindication for vaccination,
7. Not suitable for inclusion or is unlikely to comply with the protocol in the opinion of the investigator(s).

Ages: 5 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 773 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital Universitario Nuestra Señora de la Alta Gracia, Santo Domingo, Dominican Republic
- Panama (3):
  - Cevaxin Vaccination Center, David
  - Cevaxin Vaccination Center, La Chorrera
  - Cevaxin Vaccination Center, Panama City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bandyopadhyay AS, Gast C, Rivera L, Saez-Llorens X, Oberste MS, Weldon WC, Modlin J, Clemens R, Costa Clemens SA, Jimeno J, Ruttimann R. Safety and immunogenicity of inactivated poliovirus vaccine schedules for the post-eradication era: a randomised open-label, multicentre, phase 3, non-inferiority trial. Lancet Infect Dis. 2021 Apr;21(4):559-568. doi: 10.1016/S1473-3099(20)30555-7. Epub 2020 Oct 23. PMID 33284114

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - 3 Doses IPV IM: 3 doses IPV IM at 10, 14 & 36 weeks of age incl. blood sampling at 10, 14, 18 & 40 weeks.
  IPV: Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
- Group B - 2 Doses IPV IM: 2 doses IPV IM at 14 & 36 weeks of age incl. blood sampling at 14, 18, 36 & 40 weeks.
  IPV: Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
- Group C - 3 Doses f-IPV: 3 doses f-IPV ID at 10, 14 & 36 weeks of age incl. blood sampling at 10, 14, 18 & 40 weeks.
  f-IPV: Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
- Group D - 2 Doses f-IPV ID: 2 doses f-IPV ID at 14 & 36 weeks of age incl. blood sampling at 14, 18, 36 & 40 weeks.
  f-IPV: Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
Period: Overall Study
Arm/Group | Group A - 3 Doses IPV IM | Group B - 2 Doses IPV IM | Group C - 3 Doses f-IPV | Group D - 2 Doses f-IPV ID
Started | 200 | 178 | 178 | 217
Completed | 186 | 168 | 166 | 203
Not Completed | 14 | 10 | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 200 | 178 | 178 | 217 | 773
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 200 | 178 | 178 | 217 | 773
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 92 | 82 | 105 | 372
  Male | 107 | 86 | 96 | 112 | 401
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 1 | 7 | 3 | 15
  Hispanic | 105 | 108 | 101 | 132 | 446
  Latin American | 88 | 69 | 68 | 78 | 303
  White / Caucasian | 3 | 0 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Panama | 112 | 82 | 93 | 100 | 387
  Dominican Republic | 88 | 96 | 85 | 117 | 386

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Non-inferiority of 2 Doses f-IPV ID vs 2 Doses IPV IM
Description: To determine if the seroconversion rate of a 2-dose intradermally administered fractional-dose inactivated poliovirus vaccine (f-IPV) regimen administered at 14 and 36 weeks of age is non-inferior to that of a 2-dose intramuscularly administered inactivated poliovirus vaccine (IPV) regimen administered at 14 and 36 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the last dose
Population: Per Protocol Population (692 subjects) is used for this assessment. The participants flow includes the Intended to Treat population (773 subjects).
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group B | Group D
Number analyzed (Participants) | 159 | 195
percentage of seroconversion
  Serotype 1 | 98.1 [94.6 to 99.6] | 95.9 [92.1 to 98.2]
  Serotype 2 | 98.7 [95.5 to 99.8] | 97.9 [94.8 to 99.4]
Statistical Analysis 1: Comparison: Group B vs Group D; The group sizes are chosen to provide ≥ 80% power for each of the primary objectives, for the individual statistical tests of each serotype, as well as across both serotypes simultaneously. Power of ≥80% is also available for all secondary objectives, except for the comparison of the f-IPV regimen administered at weeks 14 and 36 to the 3-dose IPV regimen, which has power of 62% for individual serotypes, and 39% for the combined serotypes; Test type: Non-Inferiority — All non-inferiority comparisons of seroconversion rates will be made utilizing the lower bound of two-sided score-based confidence intervals (α = 0.05) with non-inferiority margin 10%; p = 0.05, t-test, 1 sided

2. Primary Outcome: Seroconversion Non-inferiority of 2 Doses IPV IM vs 3 Doses IPV IM
Description: To determine if the seroconversion rate of a 2-dose IPV regimen administered at 14 and 36 weeks of age is non-inferior to that of a 3-dose IPV regimen administered at 10, 14, and 36 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the last dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group A | Group B
Number analyzed (Participants) | 159 | 178
percentage of seroconversion
  Serotype 1 | 100 [97.9 to 100] | 98.1 [94.6 to 99.6]
  Serotype 2 | 100 [97.9 to 100] | 98.7 [95.5 to 99.8]
Statistical Analysis 1: Comparison: Group A vs Group B; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided

3. Primary Outcome: Seroconversion Non-inferiority of 2 Doses f-IPV ID vs 3 Doses f-IPV ID
Description: To determine if the seroconversion rate of a 2-dose f-IPV regimen administered at 14 and 36 weeks of age is non-inferior to that of a 3-dose f-IPV regimen administered at 10, 14, and 36 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the last dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group C | Group D
Number analyzed (Participants) | 160 | 195
percentage of seroconversion
  Serotype 1 | 98.8 [95.6 to 98.8] | 95.9 [92.1 to 98.2]
  Serotype 2 | 100 [97.7 to 100] | 97.9 [94.8 to 99.4]
Statistical Analysis 1: Comparison: Group C vs Group D; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Seroconversion Superiority of 2 Doses IPV IM at Different Schedules
Description: To determine if the seroconversion rate of a 2-dose IPV regimen administered at 14 and 36 weeks of age is superior to that of a 2-dose IPV regimen administered at 10 and 14 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the second dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group A | Group B
Number analyzed (Participants) | 180 | 159
percentage of seroconversion
  Serotype 1 | 95.6 [94.6 to 99.6] | 98.1 [94.6 to 99.6]
  Serotype 2 | 88.9 [83.4 to 93.1] | 98.7 [95.5 to 99.8]
Statistical Analysis 1: Comparison: Group A vs Group B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0001, Fisher Exact

5. Secondary Outcome: Seroconversion Superiority of 2 Dose f-IPV ID at Different Schedules
Description: To determine if the seroconversion rate of a 2-dose f-IPV regimen administered at 14 and 36 weeks of age is superior to that of a 2-dose f-IPV regimen administered at 10 and 14 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the second dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group C | Group D
Number analyzed (Participants) | 161 | 195
percentage of seroconversion
  Serotype 1 | 83.2 [76.5 to 88.6] | 95.9 [92.1 to 98.2]
  Serotype 2 | 83.9 [77.2 to 89.2] | 97.9 [94.8 to 99.4]
Statistical Analysis 1: Comparison: Group C vs Group D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0001, Fisher Exact

6. Secondary Outcome: Seroconversion Non-inferiority of 2 Dose f-IPV ID vs 3 Dose IPV IM
Description: To determine if the seroconversion rate of a 2-dose f-IPV regimen administered at 14 and 36 weeks of age is non-inferior to that of a 3-dose IPV regimen administered at 10, 14, and 36 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the last dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group A | Group D
Number analyzed (Participants) | 178 | 195
percentage of seroconversion
  Serotype 1 | 100 [97.9 to 100] | 95.9 [92.1 to 98.2]
  Serotype 2 | 100 [97.9 to 100] | 97.9 [94.8 to 99.4]
Statistical Analysis 1: Comparison: Group A vs Group D; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided

7. Secondary Outcome: Seroconversion Non Inferiority of 3 Doses f-IPV ID vs 3 Doses IPV IM
Description: To determine if the seroconversion rate of a 3-dose f-IPV regimen administered at 10, 14, and 36 weeks of age is non-inferior to that of a 3-dose IPV regimen also administered at 10, 14, and 36 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the last dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group A | Group C
Number analyzed (Participants) | 178 | 160
percentage of seroconversion
  Serotype 1 | 100 [97.9 to 100] | 98.8 [95.6 to 99.8]
  Serotype 2 | 100 [97.9 to 100] | 100 [97.7 to 100]
Statistical Analysis 1: Comparison: Group A vs Group C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided

8. Secondary Outcome: Seroconversion Non Inferiority of 3 Doses f-IPV ID vs 2 Doses IPV IM
Description: To determine if the seroconversion rate to a 3-dose regimen of f-IPV administered at 10, 14, and 36 weeks of age is non-inferior to that of a 2-dose IPV regimen administered at 14 and 36 weeks of age for poliovirus serotypes 1 and 2.
Time Frame: To be assessed 4 weeks after the last dose
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: percentage of seroconversion
Arm/Group | Group B | Group C
Number analyzed (Participants) | 159 | 160
percentage of seroconversion
  Serotype 1 | 98.1 [94.6 to 99.6] | 98.8 [95.6 to 99.8]
  Serotype 2 | 98.7 [95.5 to 99.8] | 100 [97.7 to 100]
Statistical Analysis 1: Comparison: Group B vs Group C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.05, t-test, 2 sided

9. Secondary Outcome: Number of Participants Experiencing SAEs, IMEs and/or Severe Local Reactions
Description: To assess the safety of each vaccine (IPV and f-IPV) as measured by the number of subjects experiencing serious adverse events (SAEs), important medical events (IMEs) and/or severe local reactions. This assessments is done in the Total Vaccinated Population (744 subjects).
Time Frame: 9 months
Population: Total Vaccinated Population (744 subjects) is used for safety analysis. The participants flow indicate the Intended To Treat population (773 subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 195 | 172 | 170 | 207
Participants
  SAE | 10 | 6 | 7 | 9
  IME | 4 | 0 | 2 | 2
  SLR | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Description: The Total Vaccinated Population (744 subjects) was used for safety analysis.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 1/195 | 0/172 | 0/170 | 0/207
Serious Adverse Events (participants affected / at risk) | 12/195 | 7/172 | 9/170 | 9/207
Other Adverse Events (participants affected / at risk) | 7/195 | 0/172 | 4/170 | 2/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=195) | Group B (N=172) | Group C (N=170) | Group D (N=207)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 4 (5) | 2 (2)
Bronchiolitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose-6-Phosphate Dehydrogenase Deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cow milk intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=195) | Group B (N=172) | Group C (N=170) | Group D (N=207)
Bronchiolitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cow milk intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03239496/Prot_SAP_000.pdf